CLINICAL TRIAL: NCT02315690
Title: Evaluating the Effectiveness and Feasibility of Reactive Focal Mass Drug Administration vs. Reactive Case Detection as a Community Level Intervention in Response to a Passively Identified Index Malaria Case in Swaziland
Brief Title: Evaluation of Reactive Focal Mass Drug Administration for Malaria Elimination in Swaziland
Acronym: fMDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ministry of Health, Swaziland (Other Government); Clinton Health Access Initiative, Eswatini (Unknown); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swaziland fMDA
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Malaria
Keywords: malaria, Swaziland, reactive case detection, focal mass drug administration
MeSH Terms: conditions — Malaria | interventions — Mass Screening; Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reactive case detection (RACD) (Active Comparator): Individuals in RACD Target Areas will be tested by RDT (rapid diagnostic test) and if positive, taken to the nearest health facility for treatment with artemether-lumefantrine per national policy.
  Interventions: Procedure: reactive case detection
- Reactive focal mass drug administration (fMDA) (Experimental): In the fMDA arm, all individuals in the Target Area will receive dihydroartemisinin-piperaquine (DHAp) once daily for 3 days with the first dose taken no later than 5 weeks from the index case presentation (goal within one week).
  Interventions: Drug: dihydroartemisinin-piperaquine (DHAp)

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine (DHAp) — In the fMDA arm, all individuals in the target area will receive dihydroartemisinin-piperaquine (DHAp) once daily for 3 days with the first dose taken no later than 5 weeks from the index case presentation (goal within one week).
  Other Names: Eurartesim
  Arms: Reactive focal mass drug administration (fMDA)
Procedure: reactive case detection — Individuals in RACD target areas will be tested by RDT and if positive will be taken to the nearest health facility for treatment as per program operating procedures.
  Other Names: screen and treat; test and treat
  Arms: Reactive case detection (RACD)

SUMMARY:
This is a cluster randomised controlled trial comparing the impact of two community based malaria interventions: reactive case detection (RACD) vs reactive targeted presumptive treatment (focal mass drug administration, fMDA) on the incidence of malaria in Swaziland.

DETAILED DESCRIPTION:
Title Evaluating the effectiveness and feasibility of reactive focal mass drug administration (fMDA) vs. reactive case detection (RACD) as a community level intervention in response to a passively identified index malaria case in Swaziland

Study design Cluster randomised controlled trial

Aims

Primary aim: To compare the impact of fMDA versus RACD on malaria incidence.

Secondary aims

Effectiveness:

1. To compare the impact of fMDA versus RACD on seroprevalence.
2. To compare the impact of fMDA versus RACD on prevalence of infection.

Feasibility:

1. To evaluate the safety of fMDA.
2. To measure the adherence of DHAp using a modified DOT regimen.
3. To determine the feasibility of reaching 80% coverage for fMDA.
4. To compare the acceptability of fMDA.
5. To compare the costs and cost-effectiveness of fMDA versus RACD.

Study site Eastern endemic region of Swaziland, a very low endemic malaria elimination setting. A total of 287 health facilities and their catchment areas are located in this area.

Time frame September 2015 - August 2017

Cluster or unit of randomisation At-risk localities will be randomized to either fMDA or RACD using a block stratified randomization based on risk rank and population

Target area Individuals residing within 200 m (fMDA arm) or 500 m (RACD arm) of an index case detected in passive surveillance, individuals residing immediately beyond 200 m in the fMDA arm will be included if a minimum of 30 individuals are not enrolled within 200 m.

Intervention All individuals residing in study localities will receive vector control preventative measures as per program. In the fMDA arm, all individuals in the target area will receive dihydroartemisinin-piperaquine (DHAp) once daily for 3 days with the first dose taken no later than 5 weeks from the index case presentation (goal within one week). Individuals in RACD target areas will be tested by RDT and taken to the nearest health facility for treatment as per program operating procedures.

Evaluation methods The primary outcome measure of incidence will be obtained through routine surveillance data.

Secondary outcomes of effectiveness will be measured at study conclusion by collecting a dried blood spot (DBS) from all residents in target areas in both arms. Prevalence of infection will be measured by loop-mediated isothermal amplification (LAMP) and seroprevalence measured by quantifying markers of recent malaria exposure.

Secondary outcomes of feasibility will be measured as follows:

1. Safety: number of serious adverse events deemed possibly, probably, or definitely related to DHAp.
2. Adherence: proportion of individuals who completed three days of therapy among all individuals initiated on DHAp in the fMDA arm, assessed by pill count.
3. Coverage: proportion of individuals residing within 200m (fMDA localities) or 500m (RACD localities) of an index case who consented to participate and who completed the initial procedures for their study arm (initial dose of DHAp in the fMDA arm or finger prick for RDT in the RACD arm).
4. Acceptability: proportion of eligible individuals refusing to take part in the study and a qualitative assessment of a subset of individuals in the fMDA arm.
5. Cost: cost per index case-level intervention and cost per case averted.

Sample size The sample size is based on the number of study localities that experienced at least one incident case of malaria in the previous season. Within 77 randomized localities, we expect that 63 localities will have an incident case of malaria and receive an intervention. For the primary objective, we hypothesize that mFDA will be more effective than RACD. At the current sample size, the study is powered to detect a difference in cumulative incidence if incidence in the fMDA arm is reduced 50% compared to the RACD arm. Incidence will be measured at the locality level and among the at-risk population, or all individuals in an enumeration area (EA) where at least one case was identified (expected to be approximately 55,928 individuals among a total study population of 211,189, or a harmonic mean of 656 per locality (41,328 effective population)). Secondary outcomes of seroprevalence and prevalence will be measured on individuals residing in target areas (total N=5,400) with a harmonic mean of 60 persons receiving intervention per locality (3,780 effective population).

Primary outcome Incidence of malaria cases

Secondary outcomes

1. Seroprevalence by ELISA
2. Prevalence of infection
3. Coverage of the intervention: proportion of the target population that receives a finger prick in the RACD arm and receives an initial dose of DHAp in the TPE arm (intention to treat analysis).
4. Adherence to DHAp in TPE arm.
5. Safety of DHAp
6. Acceptance
7. Cost per intervention episode, per case averted

ELIGIBILITY:
RACD Inclusion Criteria:

* Index case resides in study locality
* All non-index cases that reside or spent at least one night in the Target Area in the past 5 weeks
* Non-index case resides within 200 meters of index case unless study team was not able to recruit 30 individuals by 3rd visit, in which case non-index case individuals may reside up to 500 meters from index case
* Provide informed consent

RACD Exclusion Criteria:

* Refusal to participate
* Target Area overlaps with prior RACD Target Area from within the past 5 weeks

fMDA Inclusion Criteria:

* Index case resides in study locality
* All non-index cases that reside or have spent at least one night in the Target Area in the past 5 weeks
* Non-index case resides within 200 meters of index case unless study team was not able to recruit 30 individuals by 3rd visit, in which case non-index case individuals may reside up to 500 meters from index case
* Provide informed consent

fMDA Exclusion Criteria:

* Refusal to participate
* Temperature > 38.0⁰C, report of fever in the past 48 hours, or other illness (will be referred to the nearest health facility for further evaluation)
* fMDA Target Area overlaps with prior Target Area within the past 8 weeks
* For fMDA specifically (though still eligible for follow-up blood survey):

  * Pregnancy, breastfeeding, and women who have had menarche but no menses in the past 4 weeks
  * Children less than 6 months of age or <5 kg
  * Known allergy or history of adverse reaction to DP (still eligible for f/u blood surveys)
  * Already taken 2 courses of DP in the past year or taken 1 course within the past 2 months
  * Moderate or severe renal or hepatic insufficiency
  * Currently with severe malaria
  * Family history of sudden death or of congenital prolongation of the QTc (correct QT interval) interval.
  * Known congenital prolongation of the QTc-interval or any clinical condition known to prolong the QTc interval.
  * History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia. Any predisposing cardiac conditions for arrhythmia such as severe hypertension, left ventricular hypertrophy (including hypertrophic cardiomyopathy) or congestive cardiac failure accompanied by reduced left ventricle ejection fraction.
  * Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia (including vomiting in child)
  * Taking medicinal products that are known to prolong the QTc interval. See note for list of drugs.
  * Recent treatment with medicinal products known to prolong the QTc interval that may still be circulating at the time that Eurartesim is commenced (e.g. mefloquine, halofantrine, lumefantrine, chloroquine, quinine and other antimalarial agents) taking into account their elimination half-life

NOTE: Medicinal products that are known to prolong the QTc interval include:

* Antiarrhythmics (e.g. amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol).
* Neuroleptics (e.g. phenothiazines, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide, or thioridazine), antidepressive agents.
* Certain antimicrobial agents, including agents of the following classes: - macrolides (e.g. erythromycin, clarithromycin), - fluoroquinolones (e.g. moxifloxacin, sparfloxacin), - imidazole and triazole antifungal agents, - and also pentamidine and saquinavir.
* Certain non-sedating antihistamines (e.g. terfenadine, astemizole, mizolastine).
* Cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria cases | 2 years
  Cumulative incidence of malaria cases by locality

SECONDARY OUTCOMES:
Seroprevalence | during end line survey after intervention data collection completed
  Prevalence of antibody response to markers of recent malaria exposure in target areas
Prevalence | during end line survey after intervention data collection completed
  Prevalence of infection by loop mediated isothermal amplification (LAMP) in target areas
Coverage | 2 years
  Proportion of persons residing within approximately 200 m of the index case who consented to participate in the study and who completed the initial procedures for their study arm (finger prick for RDT (rapid diagnostic test) in the RACD arm, initial dose of DHAp in the fMDA arm)
Adherence | 2 years
  Proportion of persons who completed 3 days of therapy among all individuals initiated on fMDA as assessed by pill count in the first intervention per study locality
Safety related to DHAp | 2 years
  Number of participants experiencing serious adverse events (SAEs) deemed possibly, probably, or definitely related to DHAp
Acceptability | 2 years
  Qualitative assessment among individuals residing in target areas and with surveillance agents.
Cost | 2 years
  Cost per index case-level intervention, cost per case averted, collected in 10 RACD and 10 fMDA events.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Hsiang, MD, Principal Investigator — UTSW, UCSF
Locations (1):
- Swaziland Ministry of Health, Mbabane, Eswatini

REFERENCES:
- [Background] Hsiang MS, Hwang J, Kunene S, Drakeley C, Kandula D, Novotny J, Parizo J, Jensen T, Tong M, Kemere J, Dlamini S, Moonen B, Angov E, Dutta S, Ockenhouse C, Dorsey G, Greenhouse B. Surveillance for malaria elimination in Swaziland: a national cross-sectional study using pooled PCR and serology. PLoS One. 2012;7(1):e29550. doi: 10.1371/journal.pone.0029550. Epub 2012 Jan 6. PMID 22238621
- [Background] Sturrock HJ, Novotny JM, Kunene S, Dlamini S, Zulu Z, Cohen JM, Hsiang MS, Greenhouse B, Gosling RD. Reactive case detection for malaria elimination: real-life experience from an ongoing program in Swaziland. PLoS One. 2013 May 20;8(5):e63830. doi: 10.1371/journal.pone.0063830. Print 2013. PMID 23700437
- [Background] Zani B, Gathu M, Donegan S, Olliaro PL, Sinclair D. Dihydroartemisinin-piperaquine for treating uncomplicated Plasmodium falciparum malaria. Cochrane Database Syst Rev. 2014 Jan 20;2014(1):CD010927. doi: 10.1002/14651858.CD010927. PMID 24443033
- [Background] Lwin KM, Phyo AP, Tarning J, Hanpithakpong W, Ashley EA, Lee SJ, Cheah P, Singhasivanon P, White NJ, Lindegardh N, Nosten F. Randomized, double-blind, placebo-controlled trial of monthly versus bimonthly dihydroartemisinin-piperaquine chemoprevention in adults at high risk of malaria. Antimicrob Agents Chemother. 2012 Mar;56(3):1571-7. doi: 10.1128/AAC.05877-11. Epub 2012 Jan 17. PMID 22252804
- [Background] Nankabirwa JI, Wandera B, Amuge P, Kiwanuka N, Dorsey G, Rosenthal PJ, Brooker SJ, Staedke SG, Kamya MR. Impact of intermittent preventive treatment with dihydroartemisinin-piperaquine on malaria in Ugandan schoolchildren: a randomized, placebo-controlled trial. Clin Infect Dis. 2014 May;58(10):1404-12. doi: 10.1093/cid/ciu150. Epub 2014 Mar 12. PMID 24621953
- [Background] Hsiang MS, Hwang J, Tao AR, Liu Y, Bennett A, Shanks GD, Cao J, Kachur SP, Feachem RG, Gosling RD, Gao Q. Mass drug administration for the control and elimination of Plasmodium vivax malaria: an ecological study from Jiangsu province, China. Malar J. 2013 Nov 1;12:383. doi: 10.1186/1475-2875-12-383. PMID 24175930
- [Derived] Vilakati S, Mngadi N, Benjamin-Chung J, Dlamini N, Dufour MK, Whittemore B, Bhangu K, Prach LM, Baltzell K, Nhlabathi N, Malambe C, Dlamini B, Helb D, Greenhouse B, Maphalala G, Pindolia D, Kalungero M, Tesfa G, Gosling R, Ntshalintshali N, Kunene S, Hsiang MS. Effectiveness and safety of reactive focal mass drug administration (rfMDA) using dihydroartemisinin-piperaquine to reduce malaria transmission in the very low-endemic setting of Eswatini: a pragmatic cluster randomised controlled trial. BMJ Glob Health. 2021 Jun;6(6):e005021. doi: 10.1136/bmjgh-2021-005021. PMID 34193475

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02315690/Prot_SAP_ICF_001.pdf